CLINICAL TRIAL: NCT00553722
Title: Does Aldosterone Cause Hypertension by a Non-Renal Mechanism?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 1-Shavit
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-10

CONDITIONS: Hypertension; Dialysis; Hyperaldosteronism
Keywords: hypertension; dialysis; hyperaldosteronism
MeSH Terms: conditions — Hypertension; Hyperaldosteronism | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eplerenone (Experimental): Administer Eplerenone, 25 mg, orally twice daily for 4 weeks.
  Interventions: Drug: Eplerenone
- placebo (Placebo Comparator): Administer a placebo tablet orally twice daily for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplerenone — Administer Eplerenone, 25 mg,orally twice daily for 4 weeks.
  Arms: Eplerenone
Drug: Placebo — Administer a placebo tablet orally twice daily for 4 weeks.
  Arms: placebo

SUMMARY:
It is well known that Aldosterone (aldo) can cause hypertension (HBP). Since aldo is known to cause the kidney to retain sodium (Na) and Na retention is known to cause HBP, it has been thought that the mechanism by which aldo causes HBP is by Na retention. Recent studies have suggested that aldo has many effects in addition to its ability to cause the kidney to retain Na. To test the hypothesis that aldo can cause HBP in a manner which does not involve Na retention, we plan, in this protocol, to give Eplerenone, a specific aldo antagonist, to patients on dialysis who have HBP. A positive effect of Eplerenone to lower HBP in these patients would support this hypothesis.

DETAILED DESCRIPTION:
Background Shortly after the structure of aldosterone (aldo) was determined (1) in 1952, its effect on the kidney to cause sodium (Na) retention and potassium (K) and hydrogen ion (H) excretion were characterized (2,3). Although the ability of aldo to effect many transporting epithelia is now well known, it is this effect on the kidney to retain sodium which is felt to play an important role in Na retention to cause edema and, in some settings, hypertension (HBP).

Aldo was shown by Edelman (4) to bind to a specific receptor and then be transported into the nucleus of aldo responsive cells and subsequently lead to the production of aldo-induced proteins. The first aldo receptor antagonist )ARA(, spironolactone, has been used clinically for over 30 years in the management of edema and in the past few years a new agent Eplerenone, which is structurally similar to spironolactone, but without the side effect of gynecomastia, has come into clinical use in the USA and in Israel.

Treatment of HBP is usually directed at the cause of the HBP if it is known, for example, removal of tumors releasing catecholamines and correcting renal artery stenosis. If HBP is due to primary aldosteronism, then surgical removal of the tumor, or use of an ARA is usually effective (5,6). When the cause of the HBP is not known, traditionally called essential hypertension, therapy today frequently involves drugs that interfere with the RAS (7), but until recently the addition of an ARA was not usually included. Recently studies by Epstein and others (8,9) have shown that the addition of an ARA to the drug management of what has been considered essential HPB can further reduce HBP by over 10 mmHg, thus suggesting that the addition of an ARA to the routine tools available to treat HBP is important. Although the mechanism by which this addition of an ARA lowers HBP is not clear, the obvious suggestion is that by blocking the effect of aldo on the kidney to reabsorb Na there is an increased excretion of Na which is responsible for the lowering of HBP.

In patients with end-stage renal disease (ESRD), at the time they start dialysis HBP is common and has been attributed to volume overload or an active RAS (10). Early in the history of hemodialysis the potential for the RAS to be involved in causing HBP was unclear, but studies with saralasin (11,12), a competitive angiotensin II antagonist, clearly showed that in dialysis patients with elevated plasma renin levels the renin was involved in causing HBP by leading to the generation of angiotensin II. Although a number of other mechanisms apart from volume and angiotensin II have been considered, there is little evidence today that any, including aldo, play a regular role in causing HBP in the dialysis setting.

Because of the possibility that aldosterone may contribute to the HBP of patients on dialysis, independent of an effect on sodium excretion (since such patients excrete little urine), this protocol is designed to test this possibility by administering an ARA to patients on chronic dialysis with HBP. A positive result would strongly suggest that there is an effect to lower HBP independent of sodium excretion. Such a result would be indicative of a non-Na mechanism for ARA to lower HBP in dialysis patients, but would also suggest the possibility of ARA acting by a non-Na mechanism in lowering HBP in essential HBP.

Is hyperkalemia a concern in this protocol? Although there is evidence that aldo can facilitate potassium excretion, even in patients with renal failure (13) by increasing GI excretion, there have been several studies recently which demonstrate that spironolactone (14,15) or Eplerenone (16) can be given to renal failure/ dialysis patients without the development of hyperkalemia. Thus, it seems that these ARAs can be given to patients with chronic renal failure, including patients on dialysis, without hyperkalemia routinely developing. Nevertheless, in this protocol, plasma potassium will be regularly measured to minimize the development of hyperkalemia.

A very small study addressed this question using Spironolactone (14). Since it has been shown that Eplerenone does not cause gynecomastia in men, and many of our dialysis patients are men, we will use this drug, rather than Spironolactone, in this study.

Rational and Aims The role of aldo to cause HBP by a Na retaining mechanism is well described. Since recent studies suggest that aldo may have other mechanisms of action, this protocol will address the possibility that aldo can cause HBP by a non-Na retaining mechanism. This will be done by giving an ARA, Eplerenone, to patients with HBP on dialysis. In these patients the kidney plays no role in Na regulation. Thus, if BP falls with Eplerenone, these observations would strongly support the hypothesis than aldo can cause HBP by a non-Na retaining mechanism.

Methods We will select study participants from adult hemodialysis patients treated thrice weekly at Shaare Zedek Medical Center Dialysis Unit. Men and women will qualify for the study if they were on hemodialysis therapy for more than 3 months, have an average predialysis plasma potassium concentration less than 5.6 mEq/L at the time of enrollment and have nil or minimal urine output (<500 mL/24 h). All participating women of childbearing age will have a negative pregnancy test result before entering into the study. Additional exclusion criteria will include a known allergy to Spironolactone or Eplerenone; any acute illness; hypotension, defined as a predialysis systolic blood pressure less than 100 mm Hg; severe hypertension (predialysis systolic blood pressure >180 mm Hg and/or diastolic blood pressure >100 mm Hg); decompensated heart failure; inability to give informed consent; and noncompliance. The Institutional Review Board of Shaare Zedek Medical Center will be asked to give approval to the study protocol. All participants will give written-informed consent.

We plan on enrolling 27 patients in a prospective, randomized, double-blinded, placebo-controlled, crossover study. At study start, participants will be administered either Eplerenone, 25 mg, or a placebo tablet orally twice daily for 4 weeks. This 4-week period will be followed by a 3-week washout period. After the washout period, patients will cross over in their treatment arms for 4 more weeks. Patients administered Eplerenone for the first 4 weeks will be given placebo for the last 4 weeks, and vice versa. All patients will serve as their own controls.

Participants will receive outpatient hemodialysis 3 times a week using B. Braun CE0123 machines (B. Braun, D-34212 Meisungen, Germany). All patients will use B. Braun polysulfone membranes. To control for the effects of volume on blood pressure and the RAS, we plan to keep target postdialysis weight (dry weight) constant for each patient during the study. Dialysate sodium concentrations will be held constant at 140 mEq/L for all patients, dialysate potassium concentrations will be maintained at 2 mEq/L thru the study. We do not plan to impose additional dietary potassium restrictions beyond the usual recommendations for patients with ESRD treated with hemodialysis. We plan to make no changes to dialysate potassium concentrations or antihypertensive regimens. Because of a mandate not to alter the antihypertensive regimen, target weight, and dialysis potassium bath during the study, we will exclude patients with hypotension, severe hypertension, and hyperkalemia. To evaluate the effect of Eplerenone independent of its diuretic action, we plan to include only oliguric or anuric patients (urine output <500 mL/24 h).

We plan to determine predialysis and postdialysis weights, interdialytic weight gains (IDWGs), and systolic and diastolic blood pressures for each patient by calculating an average of 3 measurements obtained during 1 week before the administration of any study medication (baseline), during each week of placebo and Eplerenone treatment, and during the last week of the washout period. At the beginning and end of each treatment period, we plan to measure predialysis and postdialysis plasma potassium and aldosterone levels, renin activity (PRA), and, on a nondialysis day, 24-hour urine excretion of sodium, potassium, and creatinine. We plan to monitor predialysis plasma potassium concentrations weekly in all subjects. Predialysis blood samples will be obtained after cannulation of the vascular access before the start of the dialysis session. We plan to obtain postdialysis blood samples from a predialyzer blood sample port at the end of the hemodialysis session after slowing the blood pump to 50 to 100 mL/min. Shaare Zedek Medical Center Laboratory will perform all laboratory tests.

Statistical Methods Results will be presented as mean ± SD. To compare clinical and laboratory parameters, Student t-test will be used for paired samples. Linear regression and correlation will be used to assess the relationship between 2 variables. Stepwise regression will be used to identify predictors of a single variable. P less than 0.05 will be used to define statistical significance. We will perform all statistical analyses using standard software packages.

ELIGIBILITY:
Inclusion Criteria:

* We will select study participants from adult hemodialysis patients treated thrice weekly at Shaare Zedek Medical Center Dialysis Unit.
* Men and women will qualify for the study if they were on hemodialysis therapy for more than 3 months, have an average predialysis plasma potassium concentration less than 5.6 mEq/L at the time of enrollment and have nil or minimal urine output (<500 mL/24 h).
* All participating women of childbearing age will have a negative pregnancy test result before entering into the study.

Exclusion Criteria:

Exclusion criteria will include:

* A known allergy to Spironolactone or Eplerenone
* Any acute illness; hypotension, defined as a predialysis systolic blood pressure less than 100 mm Hg
* Severe hypertension (predialysis systolic blood pressure >180 mm Hg and/or diastolic blood pressure >100 mm Hg)
* Decompensated heart failure
* Inability to give informed consent; and
* Noncompliance.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2007-11; Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Significant drop in blood pressure with Eplerenone when compared to placebo. | days

CONTACTS AND LOCATIONS:
Overall Officials: Linda Shavit, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel